CLINICAL TRIAL: NCT01723488
Title: A Phase 0, Open Label, Non-Randomized, Multi-Center, Exploratory and Safety Study of [F-18]T808
Brief Title: A Phase 0, Open Label, Multi-Center, Exploratory and Safety Study of [F-18]T808
Acronym: T808
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study was terminated in anticipation of transfer of ownership to Avid Radiopharmaceuticals.
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: T808000
Record Dates: First submitted 2012-11-01; First posted 2012-11-08 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Alzheimers Disease
Keywords: AD
MeSH Terms: conditions — Alzheimer Disease | interventions — tau Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tau diagnostic (Experimental): Experimental: Tau diagnostic [F18] T808
  Interventions: Radiation: [F18] T808

INTERVENTIONS:
Radiation: [F18] T808 — Dose for normal volunteer undergoing dosimetry evaluation will not exceed 20 mCi, dose for high probability of Alzheimer's and low probability Alzheimer's undergoing brain imaging only will not exceed 10 mCi
  Other Names: Tau [F-18]T808

SUMMARY:
[F-18]T808 is being developed as a diagnostic radiopharmaceutical for PET imaging of the human brain.

DETAILED DESCRIPTION:
Siemens Molecular Imaging (SMI) is seeking to determine if [F-18]T808 might be useful as a non-invasive assessment tool in the clinical evaluation of subjects with conditions associated with tau protein aggregates, such as Alzheimer's disease. The information collected under this exploratory study will not be used for diagnostic purposes, assessments of the participant's response to therapy or for clinical management of the participants. However, this exploratory study will provide baseline information on the safety, biodistribution, and dosimetry of [F-18]T808. These data will aid in the design of future studies of [F-18]T808 in patients with Alzheimer's disease. Overall, this study will provide initial data that inform the development of [F-18]T808 as the first PET imaging agent for human tau protein related pathology.

ELIGIBILITY:
Low Probability for AD Participants (Group 1)

* Participant is of any race/gender/ethnicity who has reached his or her 55th birthday at the time of informed consent.
* Participant provides written informed consent Participant is capable of complying with study procedures
* Participant is capable of communicating with study personnel
* Participant understands and speaks English
* Participant has at least an 8th Grade education
* In the Investigator"s opinion, participant has a low probability of being currently positive for AD as determined by a Mini Mental State Examination (MMSE ≥ 28) defined in APPENDIX VI of XXX protocol
* Participant has no significant hepatic or renal disease as defined by previous medical history and lab results are within the following ranges: Total bilirubin within 2x institutional upper limits of normal AST (SGOT) ≤ 2.5 x institutional upper limits of normal ALT (SGPT) ≤ 2.5 x institutional upper limits of normal Creatinine ≤ 2x institutional upper limits of normal BUN within 2x institutional upper limits of normal

High Probability for AD Participants (Group 2)

* Participant is of any race/gender/ethnicity who has reached his or her 55th birthday at the time of informed consent.
* Participant or participant"s legally acceptable representative provides written informed consent Participant is capable of complying with study procedures
* Participant is capable of communicating with study personnel
* Participant understands and speaks English
* Participant has at least an 8th Grade education In the Investigator"s opinion, *participant has a high probability of being currently positive for AD that is determined by a Mini Mental State Examination (MMSE < 17) defined in APPENDIX VI of XXX protocol
* Participant has no significant hepatic or renal disease as defined by previous medical history, and lab results are within the following ranges: Total bilirubin within 2x institutional upper limits of normal AST (SGOT) ≤ 2.5 x institutional upper limits of normal ALT (SGPT) ≤ 2.5 x institutional upper limits of normal Creatinine ≤ 2x institutional upper limits of normal BUN within 2x institutional upper limits of normal

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
To monitor and assess the safety of IV administration of [F-18]T808 | up to15 days per patient.
  To monitor and assess the safety of IV administration of [F-18]T808 To evaluate the bio-distribution and radiation dosimetry of [F-18]T808 in participants with low probability of Alzheimer"s disease (AD) using PET/CT whole body imaging To evaluate the metabolism of [F-18]T808 in participants with low probability of AD using serial blood samples collected pre- and post-IP administration To evaluate [F-18]T808 uptake and signal/background information in brain PET/CT imaging of participants with a high probability of currently being positive for AD and age-matched participants with a low probability of currently being positive for AD

SECONDARY OUTCOMES:
To begin collection of baseline [F-18]T808 PET/CT imaging data | up to14 days per patient
  To begin collection of baseline [F-18]T808 PET/CT imaging data To gain information to improve the study design for the conduct of future trials

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Avid Radiopharmaceuticals
Locations (2):
- United States (2):
  - Research Site, Irvine, California
  - Research Site, Los Angeles, California